CLINICAL TRIAL: NCT01182402
Title: Electronic Compliance Monitoring in Opioid Substitution Treatment
Acronym: EHSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Ulrich Tacke, Kuopio University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KUH5703432
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Opiate Dependence
Keywords: opiate dependence; substitution treatment; unsupervised dosing; monitoring
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electronic compliance monitoring (Experimental): Suboxone treated patients in Kuopio city area get their unsupervised Suboxone doses in electronic compliance monitoring devices during the 4 month study.
  Interventions: Device: Compliance monitoring with electronic device

INTERVENTIONS:
Device: Compliance monitoring with electronic device — Patients get all their unsupervised substitution medication doses in electronic monitoring devices during the study. Daily dose of the drug is possible to get from the device in given time points and in the meantime device is locked.

SUMMARY:
The purpose of this study is to improve unsupervised dosing of opioid substitution medications. The aim of the study is to examine whether electronic compliance monitoring provides some advantages to patients'treatment and what kind of patients especially benefit from monitoring. We would also like to know if electronic compliance monitoring can prevent the abuse/diversion of medications and how implementing this method to wider treatment facilities succeeds.

ELIGIBILITY:
Inclusion Criteria:

* opiate dependence F11.22 according to ICD-10
* Suboxone treatment
* the duration of substitution treatment before study at least one month
* stable medication dose

Exclusion Criteria:

* unstable situation in life according to treatment staff's opinions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The effectiveness of treatment (Treatment Outcomes Profile TOP) | Every two months.
  Structured interview designed to measure the effectiveness and outcomes of opioid substitution treatment.

SECONDARY OUTCOMES:
Patients´opinions about the treatment. | Once when the study phase ends (after four months).
  Questionnaire designed for this study to explore patients' opinions on the compliance monitoring and it's effect on their treatment and abuse and/or diversion of medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Finland